CLINICAL TRIAL: NCT00257556
Title: A Prospective, Open Label, Randomised, Parallel Group, Comparative Pilot Study to Study the Efficacy and Safety of Highly Purified Menotrophin Versus Recombinant FSH (Follitropin Alfa) Administered Subcutaneously to Subfertile Female Patients Undergoing IVF Using Antagonist Downregulation
Brief Title: A Study of the Efficacy and Safety of Highly Purified Menotrophin Versus Recombinant Follitropin Alfa
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Clinical Development Support, Ferring Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FE999906 CS004 (PROSPECT); 2004-001307-35 (Registry Identifier: EudraCT)
Record Dates: First submitted 2005-11-22; First posted 2005-11-23 (Estimated); Results first posted 2010-02-26 (Estimated); Last update posted 2010-02-26 (Estimated); Status verified 2010-02

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Menotropins; follitropin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Menotrophin (Experimental)
  Interventions: Drug: Menotrophin
- Follitropin alfa (Active Comparator)
  Interventions: Drug: Follitropin alfa

INTERVENTIONS:
Drug: Menotrophin — 150 IU Menotrophin daily subcutaneous injection for a maximum of 13 days. In the event of hyperstimulation, the dose was reduced to 75 IU daily.
  Other Names: Menopur; hMG; highly purified menotrophin
  Arms: Menotrophin
Drug: Follitropin alfa — 150 IU follitropin alfa daily by subcutaneous injection for a maximum of 13 days. In the event of hyperstimulation, the dose was reduced to 75 IU daily.
  Other Names: rFSH; recombinant FSH
  Arms: Follitropin alfa

SUMMARY:
Prospective open label, randomised, parallel group, comparative pilot.

DETAILED DESCRIPTION:
Ongoing pregnancy rate, defined as positive fetal heart action 9 weeks after the first positive pregnancy test. Number/diameter of follicles, number of oocytes retrieved, number of pronuclear oocytes (referred to as zygotes or pre-embryos in the UK), quality of pronuclear stage oocytes, number of embryos transferred, quality of embryos, number of frozen embryos, endometrial thickness and morphology on day of HCG administration, estradiol levels at day of HCG administration, implantation rate, number of days stimulated with gonadotrophins and number of ampoules used, clinical pregnancy rate at 6 weeks after the first positive pregnancy test, pregnancy outcome.

ELIGIBILITY:
Female patients aged > or = 20 and < or = 35 years with a BMI of >18 and <32 kg/m2 who have received no more than two previous cycles of in vitro fertilisation (IVF) or other assisted reproductive technique (ART) and whose partners have normal sperm (according to WHO 1999 criteria).

Inclusion criteria:

* Signed informed consent;
* Subfertile premenopausal female patients eligible for IVF treatment;
* Aged >=20 and <=35 years;
* Body mass index of >18 and <32 kg/m2
* Normal endocrine assessment within the last 6 months;
* Normal pelvic ultrasound (showing two ovaries, no ovarian abnormalities and normal uterus) within the last 6 months;
* Receipt of no more than two previous cycles of IVF (or other ART);
* At least 3 consecutive ovulatory menstrual cycles of 24-35 days, and documented evidence of ovulatory cycles within the previous 12 months;
* No fertility-modifying treatment within the 3 months prior to this treatment cycle;
* Infertility attributable to or in association with either tubal factor, or unexplained causes;
* Sperm of partner classed as normal according to WHO 1999 criteria within the year prior to beginning therapy;
* Negative serum beta-HCG pregnancy test prior to beginning therapy;
* Clinically normal baseline haematology, clinical chemistry, and urinalysis parameter values, negative serum HBsAg and HIV antibody tests;
* Screening endocrine test results (estradiol, LH, FSH, progesterone, prolactin, TSH) in early follicular phase within the normal limits for the clinical laboratory.

Exclusion criteria

* Presence of any clinically relevant systemic disease(e.g. insulin- dependent diabetes mellitus);
* A history of or current endocrine disease, including polycystic ovary- like syndrome and hyperprolactinaemia;
* A history of coagulation disorders;
* Persistent ovarian cysts;
* Contraindications for the use of gonadotrophins or GnRH antagonists;
* A history of hypersensitivity to any of the constituents of the study medication or related compounds;
* Three or more previous cycles of IVF (or other ART);
* A history of alcohol abuse (more than 30 units per week on a regular basis);
* History of chemo- or radiotherapy;
* Currently breast-feeding, pregnant or with a contraindication to pregnancy;
* Diagnosed poor responders in prior IVF treatment;
* History of severe ovarian hyperstimulation syndrome (OHSS) (4 or 5) in former IVF treatment;
* Investigational drug within the 30 days prior to treatment;
* Any other condition or history that the investigator considers might increase the risk to the individual.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2005-10; Primary Completion 2008-07 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (6):
- Germany (3):
  - Gemeinschaftspraxis und Tagesklinik, Olpe 19, Dortmund
  - Universitats-Frauenklinik Heidelberg Abt. Gynakologische Endokrinologie und Fertilitatsstorungen, Voßstr. 9, Heidelberg
  - Gemeinschaftspraxis und Tagesklinik, Zingel 29, Hildesheim
- United Kingdom (3):
  - Royal Infirmary of Edinburgh, 51 Little France, Edinburgh
  - Leeds General Infirmary, Great George Street, Leeds
  - The Royal Hallamshire Hospital, University of Sheffield, Jessop Wing, Tree Root Walk, Sheffield

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Ninety (90) participants were screened and 80 participants randomized.
Groups:
- Menotrophin: Highly purified menotrophin sourced from human menopausal gonadotrophin (hMG)
- Follitropin Alfa: A genetically engineered substitute for follicle stimulating hormone (recombinant FSH (rFSH)).
Period: Overall Study
Arm/Group | Menotrophin | Follitropin Alfa
Started | 38 | 42
All Patients Treated Population | 37 (Also the safety population. One randomized patient did not receive study medication.) | 39 (Also the safety population. Three randomized patients did not receive study medication.)
Completed | 24 | 32
Not Completed | 14 | 10
Not completed — Adverse Event | 1 | 4
Not completed — Physician Decision | 6 | 0
Not completed — Did not meet hCG criterion | 3 | 0
Not completed — other reason | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Menotrophin | Follitropin Alfa | Total
Number analyzed (Participants) | 37 | 39 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 39 | 76
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 30.7 (3.45) | 30.9 (2.67) | 30.8 (3.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 39 | 76
  Male | 0 | 0 | 0
Tobacco Use [Number; unit: participants]
  Smoker | 4 | 8 | 12
  Ex-smoker | 8 | 5 | 13
  Never Smoked | 25 | 26 | 51
Body Mass Index [Mean (Standard Deviation); unit: Kilograms/Meters squared] — Body mass index (BMI) is measure of body fat based on height and weight that applies to both adult men and women
  Kilograms/Meters squared | 24.02 (3.689) | 23.81 (3.731) | 23.91 (3.687)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 74.1 (8.83) | 73.8 (9.96) | 74.0 (9.37)
Pulse [Mean (Standard Deviation); unit: beats per minute] | 75.7 (9.63) | 74.5 (9.16) | 75.1 (9.35)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 115.3 (12.50) | 116.1 (14.55) | 115.7 (13.51)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Ongoing Pregnancy
Description: Number of participants who met human chorionic gonadotrophin (hCG) criterion, received an embryo transfer, tested positive with a serum pregnancy test 11-14 days after embryo transfer and had an ongoing pregnancy (defined as positive fetal heart action) at ≥ 9 weeks after the first positive pregnancy test.
Time Frame: Approx week 13; 9 weeks or more after the 1st positive pregnancy test
Population: All patients treated population
Measure: Number; unit: participants
Arm/Group | Menotrophin | Follitropin Alfa
Number analyzed (Participants) | 37 | 39
participants | 14 | 13

2. Primary Outcome: Percentage of Participants With an Ongoing Pregnancy
Description: Percentage of participants who had an ongoing pregnancy ≥ 9 weeks after the first positive pregnancy test, as indicated by positive fetal heart action.
Time Frame: Approx week 13; 9 weeks or more after the first positive pregnancy test
Population: All patients treated population. Two menotrophin patients did not have pregnancy outcome data recorded in this timeframe but were later recorded as having live births so are included here as "YES" for ongoing pregnancy.
Measure: Number; unit: percentage of participants
Arm/Group | Menotrophin | Follitropin Alfa
Number analyzed (Participants) | 37 | 39
percentage of participants | 37.8 | 33.3
Statistical Analysis 1: Comparison: Menotrophin vs Follitropin Alfa; Test type: Superiority or Other; Mean Difference (Final Values) = -0.045, 95% CI [-0.170 to 0.260] — A two-sided 95% continuity-corrected confidence interval for the difference in percentages, based on the normal approximation

3. Secondary Outcome: Participants With Varying Numbers of Follicles That Were Greater Than or Equal to 17 Millimeters
Description: The criterion for ovulation induction was three follicles ≥ 17 mm diameter as shown by pelvic ultrasound examination. Patients were assessed by pelvic ultrasound on the morning (prior to menotrophin or follitropin alfa administration) of Day 7 and, if appropriate, every 2 days thereafter (Days 9/11/13) until the criterion was met.
Time Frame: Day 7 and, if appropriate, every 2 days thereafter (Days 9/11/13)
Population: All treated patients population
Measure: Number; unit: participants
Arm/Group | Menotrophin | Follitropin Alfa
Number analyzed (Participants) | 37 | 39
participants
  Did not meet criterion | 10 | 3
  3 follicles ≥ 17 mm in diameter | 11 | 11
  4 follicles ≥ 17 mm in diameter | 7 | 10
  5 follicles ≥ 17 mm in diameter | 2 | 10
  6 follicles ≥ 17 mm in diameter | 4 | 1
  7 follicles ≥ 17 mm in diameter | 0 | 0
  8 follicles ≥ 17 mm in diameter | 1 | 3
  9 follicles ≥ 17 mm in diameter | 0 | 0
  10 follicles ≥ 17 mm in diameter | 1 | 0
  11-14 follicles ≥ 17 mm in diameter | 0 | 0
  15 follicles ≥ 17 mm in diameter | 0 | 1
  16 follicles ≥ 17 mm in diameter | 1 | 0

4. Secondary Outcome: Participants With Varying Numbers of Oocytes Retrieved
Description: Number of participants with grouped by the number of oocytes retrieved. Oocytes were retrieved following ovulation induction by subcutaneous administration of human chorionic gonadotrophin (hCG) in the form of choriogonadotropin alfa at a dose of 250 micrograms once participants reached the criteria of at least three follicles with >= 17mm in diameter.
Time Frame: Approximately study day 15
Population: All treated patients population.
Measure: Number; unit: participants
Arm/Group | Menotrophin | Follitropin Alfa
Number analyzed (Participants) | 23 | 29
participants
  0 oocytes retrieved | 1 | 0
  1 oocyte retrieved | 1 | 1
  2 oocytes retrieved | 3 | 1
  3 oocytes retrieved | 3 | 1
  4 oocytes retrieved | 2 | 2
  5 oocytes retrieved | 2 | 5
  6 oocytes retrieved | 4 | 4
  7 oocytes retrieved | 2 | 2
  8 oocytes retrieved | 2 | 4
  9 oocytes retrieved | 2 | 2
  10 oocytes retrieved | 1 | 3
  11 oocytes retrieved | 0 | 0
  12 oocytes retrieved | 0 | 4
  13 oocytes retrieved | 0 | 1
  14 oocytes retrieved | 1 | 0
  15 oocytes retrieved | 0 | 3
  16 oocytes retrieved | 1 | 2
  17-18 oocytes retrieved | 0 | 0
  19 oocytes retrieved | 1 | 2
  20 oocytes retrieved | 0 | 0
  21 oocytes retrieved | 1 | 0
  22 oocytes retrieved | 0 | 0
  23 oocytes retrieved | 0 | 1

5. Secondary Outcome: Participants With Varying Numbers of Pronuclear Stage Oocytes
Description: Number of participants with various groupings of pronuclear oocytes retrieved 16-20 hours after insemination.
Time Frame: Approximately study day 15
Population: All patients treated population
Measure: Number; unit: participants
Arm/Group | Menotrophin | Follitropin Alfa
Number analyzed (Participants) | 25 | 35
participants
  1 pronuclear stage oocyte | 1 | 0
  2 pronuclear stage oocytes | 8 | 6
  3 pronuclear stage oocytes | 1 | 3
  4 pronuclear stage oocytes | 2 | 7
  5 pronuclear stage oocytes | 4 | 7
  6 pronuclear stage oocytes | 1 | 0
  7 pronuclear stage oocytes | 2 | 2
  8 pronuclear stage oocytes | 2 | 2
  9 pronuclear stage oocytes | 1 | 1
  10 pronuclear stage oocytes | 1 | 1
  11 pronuclear stage oocytes | 2 | 0
  12 pronuclear stage oocytes | 0 | 4
  13 pronuclear stage oocytes | 0 | 1
  14-16 pronuclear stage oocytes | 0 | 0
  17 pronuclear stage oocytes | 0 | 1

6. Secondary Outcome: Participants With Varying Numbers of Embryos Transferred
Description: Number of participants with various categories of numbers of embryos transferred.
Time Frame: Approximately study day 17
Population: All patients treated population
Measure: Number; unit: participants
Arm/Group | Menotrophin | Follitropin Alfa
Number analyzed (Participants) | 24 | 33
participants
  0 embryos transferred | 0 | 1
  1 embryo transferred | 3 | 1
  2 embryos transferred | 21 | 28
  3 embryos transferred | 0 | 3

7. Secondary Outcome: Participants With Varying Numbers of Embryos Frozen
Description: Number of participants with different categories of number of embryos frozen.
Time Frame: Approximately study day 17
Population: All patients treated population
Measure: Number; unit: participants
Arm/Group | Menotrophin | Follitropin Alfa
Number analyzed (Participants) | 24 | 33
participants
  0 embryos frozen | 16 | 22
  1 embryo frozen | 1 | 0
  2 embryos frozen | 2 | 1
  3 embryos frozen | 1 | 4
  4 embryos frozen | 4 | 2
  5 embryos frozen | 0 | 2
  6-8 embryos frozen | 0 | 0
  9 embryos frozen | 0 | 1
  10 embryos frozen | 0 | 1

8. Secondary Outcome: Mean Number of Days Stimulated With Gonadotrophins
Description: Number of days stimulated with study drug until participant met the criteria for ovulation induction. Ovulation induction criteria is three follicles greater than or equal to 17 mm diameter as shown by pelvic ultrasound examination.
Time Frame: study days 1 - 13
Population: All patients treated population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Menotrophin | Follitropin Alfa
Number analyzed (Participants) | 37 | 39
days | 9.2 (1.71) | 8.9 (1.07)

9. Secondary Outcome: Pregnancy Outcomes
Description: Long term follow-up to determine the outcome of the pregnancy.
Time Frame: Approximately 10 months
Population: All patients treated population
Measure: Number; unit: participants
Arm/Group | Menotrophin | Follitropin Alfa
Number analyzed (Participants) | 17 | 17
participants
  Miscarriage | 4 | 4
  Pre-term: 1 live birth | 1 | 1
  Pre-term: 2 live births | 2 | 3
  Pre-term stillbirth | 0 | 1
  Full term: 1 live birth | 7 | 6
  Full term: 2 live births | 3 | 2

10. Secondary Outcome: Mean Endometrial Thickness
Description: Measurement performed on day of human chorionic gonadotrophin (hCG) administration/ovulation induction.
Time Frame: Day 7 or 9 or 11 or 13
Population: All patients treated population
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Menotrophin | Follitropin Alfa
Number analyzed (Participants) | 27 | 38
millimeters | 11.7 (2.73) | 11.0 (2.31)

11. Secondary Outcome: Mean Estradiol Level
Description: Measurement on day of human chorionic gonadotrophin (hCG) administration / ovulation induction.
Time Frame: Day 7 or 9 or 11 or 13
Population: All patient treated population
Measure: Mean (Standard Deviation); unit: picomoles / liter
Arm/Group | Menotrophin | Follitropin Alfa
Number analyzed (Participants) | 27 | 38
picomoles / liter | 6706.6 (4109.26) | 6268.3 (4132.11)

ADVERSE EVENTS:
Description: The 'all patients treated' population is the same as the safety population in this study.
Arm/Group | Menotrophin | Follitropin Alfa
Serious Adverse Events (participants affected / at risk) | 4/37 | 9/39
Other Adverse Events (participants affected / at risk) | 18/37 | 21/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Menotrophin (N=37) | Follitropin Alfa (N=39)
Abdominal Pain (Gastrointestinal disorders) | 0 | 2
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 3
Abortion Imminent (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Ovarian Hyperstimulation Syndrome (Reproductive system and breast disorders) | 2 | 3
Uterine Haemorrhage (Reproductive system and breast disorders) | 0 | 1
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Menotrophin (N=37) | Follitropin Alfa (N=39)
Abdominal Distension (Gastrointestinal disorders) | 1 | 4
Abdominal Pain (Gastrointestinal disorders) | 0 | 2
Abdominal Pain Lower (Gastrointestinal disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3
Injection Site Bruising (General disorders) | 3 | 2
Injection Site Erythema (General disorders) | 6 | 4
Injection Site Haemorrhage (General disorders) | 0 | 3
Injection Site Pruritus (General disorders) | 7 | 2
Injection Site Rash (General disorders) | 0 | 2
Injection Site Swelling (General disorders) | 4 | 4
Nasopharyngitis (Infections and infestations) | 2 | 0
Dizziness (Nervous system disorders) | 1 | 2
Headache (Nervous system disorders) | 1 | 6
Breast Tenderness (Reproductive system and breast disorders) | 1 | 3
Ovarian Hyperstimulation Syndrome (Reproductive system and breast disorders) | 2 | 4
Vaginal Haemorrhage (Reproductive system and breast disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Skin Reaction (Skin and subcutaneous tissue disorders) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restiction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript.